CLINICAL TRIAL: NCT05448677
Title: Ezurpimtrostat Autophagy Inhibitor in Association With Atezolizumab-Bevacizumab in First Line Treatment of Unresectable Hepatocellular Carcinoma, a Phase 2b Randomized Trial
Brief Title: Ezurpimtrostat Autophagy Inhibitor in Association With Atezolizumab-Bevacizumab in First Line Treatment of Unresectable Hepatocellular Carcinoma
Acronym: ABE-LIVER
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study terminated due to recruitement issues
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Genoscience Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 38RC21.0434
Record Dates: First submitted 2022-06-27; First posted 2022-07-07 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — atezolizumab; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Ezurpimtrostat+Atezolizumab-Bevacizumab
  Interventions: Drug: Ezurpimtrostat; Drug: Atezolizumab; Drug: Bevacizumab
- Control (Active Comparator): Atezolizumab-Bevacizumab
  Interventions: Drug: Atezolizumab; Drug: Bevacizumab

INTERVENTIONS:
Drug: Ezurpimtrostat — Patients in the experimental arm will be instructed to take their assigned oral dose every day.
  Arms: Experimental
Drug: Atezolizumab — Atezolizumab will be administered by IV infusion at a fixed dose of 1200 mg on Day 1 of each 21-days cycle
Drug: Bevacizumab — Bevacizumab will be administered by IV infusion at a dose of 15 mg/kg on Day 1 of each 21-day cycle.

SUMMARY:
The study will assess the efficacy of Ezurpimtrostat in association with standard of care (Atezolizumab-Bevacizumab), compared to standard of care alone, as first line treatment in patients with unresectable hepatocellular carcinoma.The study drug which is tested is the Ezurpimtrostat in association with Atezolizumab-Bevacizumab to allow a better tumor response as well as better survival outcomes with an acceptable safety.

DETAILED DESCRIPTION:
The study is a multicentric, prospective, comparative, randomized, open-label phase 2b trial. This study will enroll 187 to 196 patients and consists of 2 parts: Safety Lead-in Phase and Expansion Phase. Initially, 3 to 12 patients will be enrolled into a Safety Lead-in Phase based on a 3 + 3 design, with the possibility of dose de-escalation, to confirm the recommended dose of Ezurpimtrostat.The randomized Expansion Phase will start after completion of Safety Lead-in Phase at the confirmed dose and will include 184 patients. Patients will be randomly assigned between experimental arm (Ezurpimtrostat + Atezolizumab-Bevacizumab) and control arm (Atezolizumab-Bevacizumab) according to a 1:1 repartition.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females ≥ 18 years of age
2. Histologically confirmed (liver biopsy within 6 previous months) and documented non resectable or metastatic HCC
3. No prior systemic therapy for advanced HCC
4. Liver tumor burden< 50% of the liver (per Investigator judgment)
5. Child-Pugh A (≤ 6) without any history of cirrhotic decompensation within the past 6 months
6. Antiviral therapy required in hepatitis B virus patients (Hepatitis B antigen positive)
7. Presence of a measurable tumor per RECIST v1.1 criteria
8. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1
9. Life expectancy ≥ 12 weeks
10. In case of cirrhosis, last esophageal varices detection by esogastroduodenal endoscopy have to be performed within last the 6 months before inclusion and since macro-vascular invasion diagnosis
11. Adequate hematologic function prior to the first dose of Ezurpimtrostat, defined as:

    11.1. Absolute neutrophils count ≥ 1500 cells/µL 11.2. Hemoglobin ≥ 9 g/dL with no transfusion within 4 weeks prior to first planned dose of Ezurpimtrostat 11.3. Platelet count > 50,000/µL with no transfusion within 2 weeks prior to first planned dose of Ezurpimtrostat
12. Adequate renal function prior to first dose, defined as 12.1. Serum creatinine < 1.5 ULN 12.2. Creatinine clearance ≥ 30 mL/min/m2 (by Cockroft-Gault equation of 24-hour urine) if creatinine ≥ 1.5 X ULN
13. Adequate hepatic function prior to first dose, defined as AST/ALT ≤ 5 X ULN
14. Women patients of childbearing potential* must have a negative blood pregnancy test at screening and baseline, and be willing to use a highly effective** contraception. The patient should be advised to continue the contraception for at least 6 months following the completion of dosing. Women with cessation for > 24 months of previously occurring menses, or women of any age who have had a hysterectomy, or have had both ovaries removed will be considered to be of non-childbearing potential
15. Male patients of reproductive potential must be willing to use one acceptable method of contraception, as judged by Investigator and Sponsor, and to refrain from donating sperm from the time of screening through at least 6 months following the completion of dose administration
16. Amenable to computed tomography (CT) with 3 or 4 phase liver or magnetic resonance imaging (MRI) of abdomen and pelvis, and CT of chest, or MRI of whole body, for initial tumor size measurements and subsequent follow-up
17. Absence of other clinically relevant abnormalities (i.e., those which do not require medical intervention) for screening laboratory test results as judged by the Investigator and Sponsor
18. Willingness and ability to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures
19. Able to understand and provide written informed consent
20. Patients covered by Health Insurance System

    * According to CTFG guideline, a woman is considered of childbearing potential (WOCBP), i.e. fertile, following menarche and until becoming post-menopausal unless permanently sterile. Permanent sterilization methods include hysterectomy, bilateral salpingectomy and bilateral oophorectomy ** Highly effective birth control method include (according to CTFG guideline): combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, transdermal); progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable); intrauterine device; intrauterine hormone-releasing system; bilateral tubal occlusion; vasectomized partner; sexual abstinence.

Exclusion Criteria:

1. Any known history of encephalopathy
2. Untreated or incompletely treated esophageal and/or gastric varices with bleeding or high-risk for bleeding
3. Known esophageal varices with recent history of bleeding (within previous 6 months)
4. Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures
5. Known fibrolamellar HCC, sarcomatoid HCC, or mixed cholangiocarcinoma and HCC
6. Chronic treatment with immunosuppressive agents (like steroids) ≤ 6 weeks prior to first planned dose of treatment
7. Major surgical procedures, open biopsy or significant traumatic injury ≤ 4 weeks prior to first dose of treatment or anticipation of major surgical procedure during the course of the trial, minor surgical procedures ≤ 1 week of first planned dose
8. Local therapy to liver within 28 days prior to initiation of study treatment or non-recovery from side effects of any such procedure
9. Any clinically significant cardiovascular condition as judged by the Investigator (such as New York Heart Association Class II or greater cardiac failure, myocardial infarction, or cerebrovascular accident within 3 months prior to Day 1 of Cycle 1, inadequately controlled arterial hypertension, unstable arrhythmia, or unstable angina)
10. Severe or uncontrolled renal condition
11. Untreated chronic hepatitis B
12. HCV infection
13. Known history of immunodeficiency diseases (e.g., active HIV)
14. Use of any prohibited concomitant medications within 14 days of the Baseline/Day 1 visit
15. Contraindication to additional liver biopsy planned between C4 and C5
16. Contraindication to iodinated contrast agent infusion or gadolinium chelate-based contrast infusion
17. Known current alcohol (> 20g/ Day in women and > 30g/ Day in men) or substance abuse
18. Malabsorption issues (e.g., gastric bypass or gastrectomy patients)
19. History of leptomeningeal disease
20. Active or history of autoimmune disease
21. History of idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography scan
22. Known active tuberculosis
23. History of malignancy other than HCC within 3 years prior to screening, with the exception of adequately treated skin basal cell carcinoma, squamous cell carcinoma or other non-melanomatous skin cancer, in-situ carcinoma of the uterine cervix, or prostate cancer that is controlled by hormone therapy (patients may continue hormone therapy while on study)
24. Pregnancy or breastfeeding, or intention of becoming pregnant during study treatment or within at least 6 months after the last dose of treatment
25. Symptomatic, untreated, or actively progressing central nervous system (CNS) metastases
26. Uncontrolled tumor-related pain
27. Uncontrolled or symptomatic hypercalcemia
28. Treatment with systemic immunostimulatory agents
29. Prior history of hypertensive crisis or hypertensive encephalopathy
30. Evidence of bleeding diathesis or significant coagulopathy
31. History of intestinal obstruction and/or clinical signs or symptoms of GI obstruction including sub-occlusive disease related to the underlying disease or requirement for routine parenteral hydration
32. Serious, non-healing or dehiscing wound, active ulcer, or untreated bone fracture
33. Metastatic disease that involves major airways or blood vessels, or centrally located mediastinal tumor masses
34. Known clinically significant or life threatening organ or systemic disease such that in the opinion of the Investigator, the significance of the disease will compromise the patient's participation in the trial
35. Known intolerance or hypersensitivity to the active ingredient or to one of the components of the study drug
36. Subject in exclusion period for another study
37. Subject who cannot be contacted in an emergency
38. All persons protected: pregnant or parturient women, breastfeeding mothers, persons deprived of liberty by judicial or administrative decision, persons subject to a legal protection measure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2022-12-15 (Actual); Primary Completion 2024-03-08 (Actual); Study Completion 2024-03-08 (Actual)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | At 36 months
  Progression-Free Survival (PFS), defined as the time from randomization to the occurrence of disease progression or death from any cause, whichever occurs first.
  Progression events will be considered based on centralized tumor response assessment according to RECIST version 1.1 and PFS analyses will be performed by the CHU Grenoble Alpes Statistics department.

SECONDARY OUTCOMES:
Objective response rate (ORR) | At 3,6,9,12 months
  Best overall objective response rate (ORR) and ORR at 3,6,9,12 months according to RECIST 1.1 and IRF-assessed tumor response according to HCC mRECIST

CONTACTS AND LOCATIONS:
Overall Officials: Gaël ROTH, MD PHD, Principal Investigator — University Hospital, Grenoble
Locations (1):
- University Hospital, Grenoble, France

IPD SHARING:
Plan to Share IPD: No